CLINICAL TRIAL: NCT06600165
Title: Intraoperative Confocal Laser Scanning Microscopy and Artificial Intelligence for Optimized Surgical Excision of Basal Cell Carcinoma
Brief Title: Intraoperative Confocal Laser Scanning Microscopy With Use of AI for Optimized Surgical Excision of Basal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Maximilian Deußing, Principal Investigator, LMU Klinikum
Other Study IDs: DFG 536381342
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ex vivo confocal microscopy — The aim is to use AI to assist surgeons in analyzing CLSM tissue slide images obtained during BCC surgeries with the aim to integrate it in real time. We plan to use AI to analyze CLSM images of BCCs and distinguish between tumor tissue, inflammatory tissue, and non-tumor/non-inflammatory tissue. This approach would provide surgeons with real-time feedback and automated image analysis, leading to a more targeted and efficient approach to tissue analysis. By improving the accuracy and speed of tissue analysis, our proposal could ultimately improve operative patient outcomes and benefit healthcare professionals.

SUMMARY:
The aim is to use AI to assist surgeons in analyzing CLSM tissue slide images obtained during BCC surgeries with the aim to integrate it in real time. We plan to use AI to analyze CLSM images of BCCs and distinguish between tumor tissue, inflammatory tissue, and non-tumor/non-inflammatory tissue. This approach would provide surgeons with real-time feedback and automated image analysis, leading to a more targeted and efficient approach to tissue analysis. By improving the accuracy and speed of tissue analysis, our proposal could ultimately improve operative patient outcomes and benefit healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Basal Cell Carcinoma

Exclusion Criteria:

* Patient unable to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Basal Cell Carcinoma undergoing biopsy or surgery
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ex vivo confocal laser scanning microscopy | 2 years
  Reaching the planned number of 1000 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic and Policlinic of Dermatology and Allergy, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No